CLINICAL TRIAL: NCT00233675
Title: A 12-Month, Open-Label, Flexible-Dosage Study to Evaluate the Safety of GABITRIL at Dosages up to 16mg/Day in Adults With Generalized Anxiety Disorder
Brief Title: Evaluate the Safety of GABITRIL in Adults With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C6671A/301/AX/US
Record Dates: First submitted 2005-09-27; First posted 2005-10-06 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: General Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Tiagabine

INTERVENTIONS:
Drug: GABITRIL (tiagabine hydrochloride; CEP-6671)

SUMMARY:
To assess the long-term safety and tolerability of tiagabine treatment in patients with generalized anxiety disorder (GAD).

ELIGIBILITY:
Not available at time of registration

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2003-08; Primary Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brown, MD, Study Director — Cephalon
Locations (28):
- United States (28):
  - Pivotal Research Center, Mesa, Arizona
  - Southwestern Research, Beverly Hills, California
  - Pharmacology Research Institut, Newport Beach, California
  - Pharmacology Research Institut, Northridge, California
  - Pacific Clinical Research Medi, Orange, California
  - Radiant Research San Diego, San Diego, California
  - Affiliated Research Institute, San Diego, California
  - Radiant Research Denver, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Clinical Neuroscience Solution, Jacksonville, Florida
  - Clinical Neuroscience Solution, West Palm Beach, Florida
  - Carman Research, Smyrna, Georgia
  - Cunningham Clinical Research, Edwardsville, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Summit Research Network Farmin, Farmington Hills, Michigan
  - CNS Research Institute, Clementon, New Jersey
  - Social Psychiatry Research Ins, Brooklyn, New York
  - Fieve Clinical Services, Inc., New York, New York
  - Medical and Behavioral, New York, New York
  - Medical Research Network, New York, New York
  - Richard Weisler, MD and Assoc, Raleigh, North Carolina
  - Summit Research Network Inc., Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - South East Health Consultants, Charleston, South Carolina
  - Claghorn-Lesem Research, Bellaire, Texas
  - Radiant Research Salt Lake, Salt Lake City, Utah
  - Comprehensive Neuroscience Of, Falls Church, Virginia
  - Summit Seattle Boren, Seattle, Washington